CLINICAL TRIAL: NCT01787422
Title: Comparison of Telemedicine Versus Traditional Practice in a University Health Center
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator has left the university
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ASUIRB1210008469
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Health Service Research on Telemedicine
Keywords: Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemedicine Visit (Experimental): Patients who are seen by use of an off-site telemedicine physician.
  Interventions: Other: Traditional versus Telemedicine office visit
- Traditional Visit (Active Comparator): Patients who are seen in followup with a traditional in-office visit.
  Interventions: Other: Traditional versus Telemedicine office visit

INTERVENTIONS:
Other: Traditional versus Telemedicine office visit

SUMMARY:
This study is to determine if telemedicine visits provide similar quality and patient/physician satisfaction as traditional office visits in a college health population.

DETAILED DESCRIPTION:
This study which is open to students at Arizona State University who require follow-up care after their visit to ASU Health Services. Patients who are seen by a Mayo Clinic physician working at the ASU Health Services are randomized to either be seen for followup at the health center with the same physician or seen at the health center by the same physician at Mayo clinic utilizing telemedicine.

After the visit, patients and the physician will fill out an patient satisfaction survey and the record will be reviewed by an independent investigator for determining quality of care by reviewing the record.

ELIGIBILITY:
Inclusion Criteria:

* Arizona State University students who require a follow-up care visit.
* ages 18 and above

Exclusion Criteria:

* patients who are medically unstable to be randomized to a telemedicine visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Quality of care score between the two groups | At the 24 hour visit
  Using a independent quality assessor, each visit whether telemedicine will give a quality score based on adequacy of care, ability to examine/determine the diagnosis based on the documented care in the record.

CONTACTS AND LOCATIONS:
Overall Officials: Allan L Markus, MD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University Health Services, Tempe, Arizona, United States